CLINICAL TRIAL: NCT01833507
Title: Relationship Between Physical Activity and Health Outcomes in Overweight and Obese Medically Complex Adults, a Randomized Trial
Brief Title: Physical Activity and Health Outcomes
Acronym: PAHO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Paul Takahashi,, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-000675
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Overweight; Obese
Keywords: increased activity; weight loss; obesity
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- self-exercise (Active Comparator): Intervention will include a video(DVD) on exercise, and 2 self-help manuals on exercise and nutrition, in addition to a journal and pedometer.
  Interventions: Behavioral: Self-Exercise
- usual care (Placebo Comparator): Participants will have full access to all of the educational materials which are available to all Mayo Clinic patients in literature racks in the individual clinics.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Self-Exercise — Behavioral Goal Setting
  Arms: self-exercise
Behavioral: Usual Care — Participants will have full access to all of the educational materials which are available to all Mayo Clinic patients in literature racks in the individual clinics. Participants will subsequently be given entry into the active intervention at the 2-month check.
  Arms: usual care

SUMMARY:
Obesity is common in adults with complex medical problems with ensuing complications afterwards. Obese patients suffer higher mortality and impaired functional status often as a result of their obesity. One primary goal to reduce both obesity and improve functional status is exercise. The investigators hypothesize that a simple exercise intervention with limited behavioral goal-setting will reduce weight and increase functional status compared to usual care. As a secondary measure, the investigators hypothesize that using this intervention will reduce hospital admissions and ER visits.

DETAILED DESCRIPTION:
We are enrolling up to 150 subjects where half will receive a pedometer and behavioral goal-setting at enrollment and half will receive a pedometer and goal-setting 2 months later. It is a 4 month study. Our aims are as follows:

Primary Aim: Determine the relationship between gait speed, grip strength and walking steps in patients randomized to a self-exercise program compared to usual care in complex medical patients.

Second Primary aim: To determine the effect of a self-exercise program compared to usual care on weight loss in complex medical patients.

Secondary Aim: Determine the relationship between the number of hospitalizations in patients randomized to a self-exercise program compared to usual care in complex medical patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be over the age of 18
2. Have a BMI over 25.0 kg/m2.
3. Have a Minnesota Medical Tiering concerning medical complexity of 3-4.

Exclusion Criteria:

1. Patients will be excluded if they have clinically documented dementia.
2. Subjects will be community dwelling and patients living in skilled nursing facilities will be excluded.
3. Subjects residing within a correctional institution will be excluded.
4. Subject is a female patient who is currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Gait, Grip and Walking | 4 months
  Determine the relationship between gait speed, grip strength and walking steps in patients randomized to a self-exercise program compared to usual care in complex medical patients.
weight loss | 4 months
  To determine the effect of a self-exercise program compared to usual care on weight loss in complex medical patients.

SECONDARY OUTCOMES:
number of hospitalizations | 4 months
  Determine the relationship between the number of hospitalizations in patients randomized to a self-exercise program compared to usual care in complex medical patients.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Y Takahashi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States